CLINICAL TRIAL: NCT04006184
Title: Venaseal Versus Ablation With Endothermal Laser or Radiofrequency for Saphenous Vein Incompetence: a Comparison of Utilization of Adjunctive Phlebectomy
Brief Title: Retrospective Review of Saphenous Vein Incompetence: Venaseal Versus Endovenous Thermal Ablation
Acronym: VALUE
Status: Completed | Type: Observational
Sponsor: Lake Washington Vascular (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: GG2019/01
Record Dates: First submitted 2019-06-29; First posted 2019-07-05 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Varicose Veins; Venous Reflux; Venous Insufficiency
Keywords: Venaseal; Symptomatic Varicose Veins
MeSH Terms: conditions — Varicose Veins; Venous Insufficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endovenous Thermal Ablation: Limbs treated with either radiofrequency ablation or endovenous laser ablation
  Interventions: Other: Chart review
- Cyanoacrylate Closure: Limbs treated with cyanoacrylate closure system
  Interventions: Other: Chart review

INTERVENTIONS:
Other: Chart review — Retrospective review of medical records at a single site with six physicians

SUMMARY:
This study is a retrospective, chart review of treatment of patients with symptomatic varicose veins. Treated limbs must have the Great Saphenous Vein and/or Small Saphenous Vein treated with either cyanoacrylate closure (VenaSeal) or Endothermal Ablation (either Radiofrequency Ablation or Endovenous Laser Ablation).

DETAILED DESCRIPTION:
This single site, retrospective, comparison study aims to review up to 400 treated limbs with symptomatic varicose veins to compare the need for/utilization of adjunctive phlebectomy performed as a concomitant or staged procedure in conjunction with either cyanoacrylate closure versus endothermal ablation of incompetent saphenous veins through 6 months of the index procedure. The overall cost of treatment for both groups will be compared.

Some of the secondary aims of this study include:

1. To assess changes in Clinical, Etiology, Anatomy, and Pathology (CEAP) clinical class after completion of treatment.
2. To assess changes in revised Venous Clinical Severity Score (rVCSS) and compare the two groups.
3. To assess the need for adjunctive therapies.
4. To record and compare retrospectively the adverse events between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Limb with saphenous vein incompetence, treated with one of the following:

   VenaSeal ™ Endovenous Laser Ablation Radiofrequency Ablation
2. CEAP Clinical Class between 2-5
3. Limb treated from October 1st, 2015-present
4. At least 2 months of follow-up post index procedure
5. Treatment of either the great saphenous vein (GSV), the small saphenous vein (SSV), or both. Treatment of accessory saphenous veins (ASV) is allowed as long as either the GSV, SSV, or both the GSV and SSV were treated as well in that limb at the index procedure.

Exclusion Criteria:

1. Limb treatment of the accessory saphenous vein (ASV) without concomitant great saphenous vein (GSV) and/or small saphenous vein (SSV) treatment
2. Limb treatment for reasons other than symptomatic varicose veins
3. Limbs without follow-up information at least 2 months following the index procedure
4. Subjects who participated in another clinical trial as part of their saphenous vein treatment
5. Investigator decision (concurrent condition that would make inclusion inappropriate, protected subject population) -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 327 limbs treated with Cyanoacrylate Closure and 327 limbs treated with Endovenous Thermal Ablation for symptomatic varicose veins and incompetence of the great or small saphenous vein, or both veins.
Sampling Method: Probability Sample
Enrollment: 547 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Adjunctive phlebectomy | Through 6 months of index procedure
  Compare need for/utilization of adjunctive phlebectomy performed as a concomitant or staged procedure
Cost of Treatment | Through six months of index procedure
  A cost analysis will be performed calculating the total cost of treatment between groups

SECONDARY OUTCOMES:
Severity of Disease | At treatment through six months of index procedure
  Assess potential change in clinical class using the Clinical, Etiology, Anatomy, and Pathology (CEAP) clinical class
Severity of Disease | At treatment through six months of index procedure
  Assess potential change in clinical severity score using the Revised Venous Clinical Severity Score (rVCSS).
Utilization of adjunctive treatments | Through six months of index procedure
  Assess utilization of adjunctive sclerotherapy, either for cosmetic or medical need
Adverse events reported during clinic visits | Though six months of index procedure
  If adverse events were reported and documented in chart, these will be collected and categorized to assess for comparison between groups

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen D Gibson, MD, Principal Investigator — Lake Washington Vascular, PLLC
Locations (1):
- Lake Washington Vascular, PLLC, Bellevue, Washington, United States

IPD SHARING:
Plan to Share IPD: No